CLINICAL TRIAL: NCT06735794
Title: Spaced iTBS: Effects on Plasticity in the Motor Cortex
Brief Title: Impact of Spaced iTBS on Plasticity in the Motor Cortex
Acronym: STEP-MC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2023/218
Record Dates: First submitted 2024-11-22; First posted 2024-12-16 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2024-10

CONDITIONS: Healthy Control Subjects
Keywords: TMS; TBS; Brain stimulation; Healthy; Control; Healthy individuals; Transcranial Magnetic Stimulation; Intermittent Theta-Burst Stimulation; Motor Cortex; Neuroplasticity; Brain plasticity; Cortical plasticity; iTBS; iTBS-c; iTBS-s; iTBS-sh; Spaced iTBS; Compressed iTBS; Sham iTBS; LTP; Long Term Potentiation; Theta-Burst Stimulation

STUDY DESIGN:
Intervention Model Description: This study will employ a randomized, single-blind cross-over design with three experimental iTBS conditions (iTBS-c, iTBS-s, and iTBS-sh).
Who Masked: Participant
Masking Description: This clinical trial is a single-blinded study. Participants will be blinded to the iTBS condition they are receiving in Visits 2-5. The individual administering iTBS (i.e., the interventionist) will not be blinded to the iTBS condition being administered. To maintain participant blinding, each of the three iTBS interventions (iTBS-c, iTBS-s, and iTBS-sh) were designed to be similar in length and structure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Compressed iTBS (Active Comparator): After completing Visits 1-2 (Screening and Calibration), participants will undergo the iTBS-c condition in a randomized order during Visits 3 to 5. iTBS-c is the active comparator.
  Interventions: Device: Compressed iTBS
- Spaced iTBS (Experimental): After completing Visits 1-2 (Screening and Calibration), participants will undergo the iTBS-s condition in a randomized order during Visits 3 to 5. iTBS-s is the experimental study intervention.
  Interventions: Device: Spaced iTBS
- Sham iTBS (Sham Comparator): After completing Visits 1-2 (Screening and Calibration), participants will undergo the iTBS-sh condition in a randomized order during Visits 3 to 5. iTBS-sh is the sham comparator.
  Interventions: Device: Sham iTBS

INTERVENTIONS:
Device: Compressed iTBS — Intermittent Theta-Burst Stimulation (iTBS) is a form of non-invasive brain stimulation that uses magnetic pulses applied to the scalp using a coil. iTBS will be used to stimulate the left motor cortex to enhance long-term potentiation (LTP)-like activity, a physiological mechanism associated with brain plasticity.
  During the intervention, the study team will conduct two pre-iTBS TMS measurements (Pre-30 and Pre-15). Participants will then complete iTBS-c (active comparator), which will be delivered unilaterally to the left motor cortex. Following iTBS-c, five post-iTBS TMS measurements (Post-0, 15, 30, 45, and 60) will be obtained. Motor evoked potentials (MEPs) will be recorded from the right APB, ADM, and FDI muscles to assess the effects of the stimulation.
  The MCF-B65, MCF-P-B65, and/or Cool-B65 A/P TMS coils will be used, alongside the MagPro R30 or the MagPro X100 TMS stimulators to deliver the intervention.
  Other Names: iTBS-c
  Arms: Compressed iTBS
Device: Spaced iTBS — Intermittent Theta-Burst Stimulation (iTBS) is a form of non-invasive brain stimulation that uses magnetic pulses applied to the scalp using a coil. iTBS will be used to stimulate the left motor cortex to enhance long-term potentiation (LTP)-like activity, a physiological mechanism associated with brain plasticity.
  During the intervention, the study team will conduct two pre-iTBS TMS measurements (Pre-30 and Pre-15). Participants will then complete iTBS-s (experimental study intervention), which will be delivered unilaterally to the left motor cortex. Following iTBS-s, five post-iTBS TMS measurements (Post-0, 15, 30, 45, and 60) will be obtained. Motor evoked potentials (MEPs) will be recorded from the right APB, ADM, and FDI muscles to assess the effects of the stimulation.
  The MCF-B65, MCF-P-B65, and/or Cool-B65 A/P TMS coils will be used, alongside the MagPro R30 or the MagPro X100 TMS stimulators to deliver the intervention.
  Other Names: iTBS-s
  Arms: Spaced iTBS
Device: Sham iTBS — Intermittent Theta-Burst Stimulation (iTBS) is a form of non-invasive brain stimulation that uses magnetic pulses applied to the scalp using a coil. iTBS will be used to stimulate the left motor cortex to enhance long-term potentiation (LTP)-like activity, a physiological mechanism associated with brain plasticity.
  During the intervention, the study team will conduct two pre-iTBS TMS measurements (Pre-30 and Pre-15). Participants will then complete iTBS-sh (sham comparator), which will be delivered unilaterally to the left motor cortex. Following iTBS-sh, five post-iTBS TMS measurements (Post-0, 15, 30, 45, and 60) will be obtained. Motor evoked potentials (MEPs) will be recorded from the right APB, ADM, and FDI muscles to assess the effects of the stimulation.
  The MCF-B65, MCF-P-B65, and/or Cool-B65 A/P TMS coils will be used, alongside the MagPro R30 or the MagPro X100 TMS stimulators to deliver the intervention.
  Other Names: iTBS-sh
  Arms: Sham iTBS

SUMMARY:
The goal of this clinical trial is to explore the effects of non-invasive brain stimulation protocols using intermittent theta-burst stimulation (iTBS) on brain plasticity in healthy, right-handed individuals aged 18 to 50 years. Brain plasticity is the brain's ability to change through growth or reorganization. iTBS is a form of transcranial magnetic stimulation (TMS), where magnetic pulses are applied to the scalp using a coil. These pulses pass through the scalp, and can alter brain activity in the area underneath the coil. Based on previous research conducted in animals and humans, researchers believe that iTBS can strengthen the connections between cells in the brain, leading to improved brain plasticity.

This trial will compare the effects of the compressed iTBS (iTBS-c) protocol, which is commonly used to treat depression, and the spaced iTBS (iTBS-s) protocol. Researchers want to find out which protocol is better able to produce changes in brain plasticity. Sham iTBS (iTBS-sh) will be used as a control to make the results of the study more reliable.

Participants will complete 5 study visits within the span of 3 months, including:

* Screening assessments to determine eligibility (Visit 1);
* Calibration iTBS session (Visit 2) to assess tolerability of brain stimulation;
* Three experimental iTBS sessions (iTBS-s, iTBS-c, and iTBS-sh) in a randomized order (Visits 3-5), each separated by at least 72 hours. During each session, the study team will stimulate the motor cortex and record the muscle activity of your hand to measure changes in brain plasticity.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is a mental illness affecting millions of individuals worldwide and in Canada, and is a leading cause of morbidity, mortality, and disability. While antidepressant medications are effective in treating MDD, their efficacy is moderate and systemic side-effects persist, such as sexual dysfunction, drowsiness, weight gain, and dry mouth. Thus, more effective treatments are needed for MDD.

Neuroimaging techniques have implicated the dysregulation of brain plasticity in depression. In particular, long-term potentiation (LTP)-like activity in the dorsolateral prefrontal cortex (DLPFC) and the motor cortex is known to be impaired in MDD. As such, transcranial magnetic stimulation (TMS)-based interventions, which aim to modify underlying cortical activity, are now established treatments of depression. Intermittent theta-burst stimulation (iTBS), a novel form of repetitive TMS approved by the US Food and Drug Administration (FDA) for the treatment of depression, delivers intermittent, high-frequency theta bursts. It has been demonstrated to induce sustained plasticity in the DLPFC and the motor cortex. Although iTBS is approved for the treatment of depression, response and remission rates for MDD are still relatively low.

Based on promising research conducted in the hippocampus of rodents, the investigators believe that modifying some parameters of the iTBS protocol may be more effective in inducing plasticity than the currently used iTBS protocol. Thus, in this trial researchers aim to optimize iTBS and its effects on cortical plasticity as a first step towards optimizing it for the treatment of depression.

The primary and secondary objectives and hypotheses of the study are as follows:

Objective 1: To compare the effect of compressed iTBS (iTBS-c) to spaced iTBS (iTBS-s) on LTP-like activity (referred to hereafter as iTBS-LTP) as measured using motor evoked potentials (MEPs) recorded from the right abductor pollicis brevis (APB), abductor digiti minimi (ADM), and first dorsal interosseous (FDI) muscles.

Hypothesis 1: iTBS-s will elicit larger iTBS-LTP post-iTBS as compared to iTBS-c.

Objective 2: To compare the effect of iTBS-c and iTBS-s on iTBS-LTP relative to iTBS-sh.

Hypothesis 2: iTBS-c and iTBS-s will elicit larger iTBS-LTP post-iTBS as compared to iTBS-sh.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or above, and less than 51 years.
2. Right handedness, assessed using the Edinburgh Handedness Inventory (EHI).
3. Sufficiently proficient in English to complete the required study assessments, as per investigator judgement.
4. Willingness and capacity to provide informed consent.
5. Willingness to comply with all study procedures.

Exclusion Criteria:

1. Age 17 years or less, or greater than 51 years, as brain plasticity is known to be affected by age.
2. Current use of any psychotropic medications (e.g. anti-depressants, anti-convulsants, anti-psychotics, etc.).
3. Contraindications to transcranial magnetic stimulation (TMS), as per investigator judgment.
4. Lifetime history of any Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnosis, assessed using the Structured Clinical Interview for DSM-5 (SCID-5), except simple phobias.
5. Left handed or ambidextrous, assessed using the EHI, to minimize the heterogeneity in cortical excitability and plasticity.
6. Self-reported history of seizures and/or other major neurological conditions, as per investigator judgement, due to the risk of seizures associated with TMS in individuals with a heightened risk.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2024-11-13 (Actual); Primary Completion 2026-02-01 (Actual); Study Completion 2026-02-01 (Actual)

PRIMARY OUTCOMES:
iTBS-LTP | Up to 3 months
  The primary outcome measure is iTBS-induced LTP (iTBS-LTP), which will be calculated at each post-iTBS time points (Post-0, Post-15, Post-30, Post-45 and Post-60).
  At each time point, the mean or median MEP amplitude will be divided by the mean or median MEP amplitude across the two pre-iTBS TMS measurements (Pre-30 and Pre-15) for the corresponding iTBS condition. This will be repeated for all three iTBS conditions to generate iTBS-LTP values at the five post-iTBS time points. Larger iTBS-LTP values are indicative of stronger plasticity following the intervention.
  This will address hypothesis 1, which examines whether iTBS-s induces stronger iTBS-LTP compared to iTBS-c, and hypothesis 2, which evaluates whether iTBS-s and iTBS-c induce stronger iTBS-LTP compared to iTBS-sh.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Berlim MT, McGirr A, Rodrigues Dos Santos N, Tremblay S, Martins R. Efficacy of theta burst stimulation (TBS) for major depression: An exploratory meta-analysis of randomized and sham-controlled trials. J Psychiatr Res. 2017 Jul;90:102-109. doi: 10.1016/j.jpsychires.2017.02.015. Epub 2017 Feb 21. PMID 28254709
- [Result] Chung SW, Hoy KE, Fitzgerald PB. Theta-burst stimulation: a new form of TMS treatment for depression? Depress Anxiety. 2015 Mar;32(3):182-92. doi: 10.1002/da.22335. Epub 2014 Nov 28. PMID 25450537
- [Result] Höflich G, Kasper S, Hufnagel A, Ruhrmann S, Möller HJ. Application of transcranial magnetic stimulation in treatment of drug-resistant major depression-a report of two cases. Human Psychopharmacology: Clinical and Experimental. 1993;8(5):361-365.
- [Result] George MS, Wassermann EM, Williams WA, Callahan A, Ketter TA, Basser P, Hallett M, Post RM. Daily repetitive transcranial magnetic stimulation (rTMS) improves mood in depression. Neuroreport. 1995 Oct 2;6(14):1853-6. doi: 10.1097/00001756-199510020-00008. PMID 8547583
- [Result] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832
- [Result] Cantone M, Bramanti A, Lanza G, Pennisi M, Bramanti P, Pennisi G, Bella R. Cortical Plasticity in Depression. ASN Neuro. 2017 May-Jun;9(3):1759091417711512. doi: 10.1177/1759091417711512. PMID 28629225
- [Result] Vignaud P, Damasceno C, Poulet E, Brunelin J. Impaired Modulation of Corticospinal Excitability in Drug-Free Patients With Major Depressive Disorder: A Theta-Burst Stimulation Study. Front Hum Neurosci. 2019 Feb 26;13:72. doi: 10.3389/fnhum.2019.00072. eCollection 2019. PMID 30863297
- [Result] Liu W, Ge T, Leng Y, Pan Z, Fan J, Yang W, Cui R. The Role of Neural Plasticity in Depression: From Hippocampus to Prefrontal Cortex. Neural Plast. 2017;2017:6871089. doi: 10.1155/2017/6871089. Epub 2017 Jan 26. PMID 28246558
- [Result] Duman RS. Pathophysiology of depression: the concept of synaptic plasticity. Eur Psychiatry. 2002 Jul;17 Suppl 3:306-10. doi: 10.1016/s0924-9338(02)00654-5. PMID 15177086